CLINICAL TRIAL: NCT00162669
Title: Phase II Study Evaluating the Efficacy of Bevacizumab (Avastin@) in Hepatocellular Carcinoma Not Amenable to Curative Treatment
Brief Title: Bevacizumab in Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGR 1123; HCC-Avastin
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma, advanced, bevacizumab, phase II, VGEF, neovascularization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neovascularization, Pathologic | interventions — Bevacizumab

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
Primary liver cancer (hepatocellular carcinoma) is the fifth most common malignant disorder, with an increasing incidence in Europe and the USA as a result of the high prevalence of hepatitis C. Most patients are not suitable for potentially curative treatment. There is no standard palliative treatment for patients with advanced hepatocellular carcinoma (HCC), as no drug has been demonstrated to be efficient in this disease in terms of survival. The use of anti-vascular agents might be a promising approach in view of the highly vascular nature of this tumor. The aim of this phase II trial is to evaluate the potential benefit of bevacizumab in terms of disease control rate, progression-free and overall survival in adult patients with advanced primary liver cancer. Bevacizumab is an angiogenesis inhibitor already successfully used in patients with colorectal and renal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven HCC or alpha-fetoprotein level > 400 ng/ml together with hypervascular tumor and cirrhosis documented by CT scan or MRI.
* HCC not amenable to curative treatment (resection, transplantation, percutaneous ablation)
* Presence of at least one dimensionally measurable target lesion with largest diameter >= 2 cm.
* No previous chemoembolization, no previous radiotherapy
* Cancer of the Liver Italian Program (CLIP) score < 4
* World Health Organization (WHO) performance status of 2 or less
* Life expectancy >= 3 months.
* Age >= 18 years.
* Adequate hematologic functions (neutrophil count, at least 1500 per cubic millimeter; platelet count, at least 75,000 per cubic millimetre; Hemoglobin, at least 8 g/dl)
* Adequate liver function (bilirubin, not more than 2 times the upper limit of normal); Adequate renal function (serum creatinine, less than 150 micromol per liter)
* Adequate coagulation function
* Written informed consent

Exclusion Criteria:

* Decompensated cirrhosis (Child-Pugh score > 7)
* CLIP score > 4
* Variceal bleeding during the previous 3 months
* Thromboembolic event during the previous 6 months
* Medical condition requiring full dose anticoagulation or anti-platelet drugs
* Abnormal cardiac function with history of ischemic heart disease in the previous 6 months, uncontrolled hypertension, unstable angina, severe cardiac arrhythmia,
* No brain metastasis, No bone metastasis only
* Previous or current malignancies at other sites
* No concomitant antitumor treatment including tamoxifen or somatostatin analogs
* Unstable systemic diseases or active uncontrolled infections.
* Patients (male and female) not using effective contraception if of reproductive potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-05

PRIMARY OUTCOMES:
The main response parameter will be the disease control rate, defined by the objective response and stable disease rate (Response Evaluation Criteria in Solid Tumors [RECIST criteria]) after two consecutive tumor evaluations during treatment.

SECONDARY OUTCOMES:
Overall survival, progression-free survival, toxicity (National Cancer Institute-Common Toxicity Criteria Version 3 [NCI-CTC V3])
Evaluation of vascular changes will be performed using Doppler ultrasound with injection of sonographic contrast agent

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BOIGE, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Boige V, Malka D, Bourredjem A, Dromain C, Baey C, Jacques N, Pignon JP, Vimond N, Bouvet-Forteau N, De Baere T, Ducreux M, Farace F. Efficacy, safety, and biomarkers of single-agent bevacizumab therapy in patients with advanced hepatocellular carcinoma. Oncologist. 2012;17(8):1063-72. doi: 10.1634/theoncologist.2011-0465. Epub 2012 Jun 15. PMID 22707516